CLINICAL TRIAL: NCT00756938
Title: A Phase III, Randomized, Open-Label, Parallel-Group, Dose-Ranging Clinical Trial to Study the Safety and Efficacy of MK954/Losartan Potassium in Pediatric Patients With Hypertension
Brief Title: Study of Losartan in Pediatric Patients With Hypertension (MK-0954-337)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0954-337; 2008_545 (Other: Merck Study Number); CTRI/2009/091/000045 (Registry Identifier: CTRI)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Losartan potassium 0.1 to 1.4 mg/kg (Experimental): Open-label losartan at starting dose of 0.1 mg/kg/day with uptitration at Weeks 3, 6, or 9 to the next highest dose level if blood pressure goal not achieved
  Interventions: Drug: losartan potassium
- Losartan potassium 0.3 to 1.4 mg/kg (Experimental): Open-label losartan at starting dose of 0.3 mg/kg/day with uptitration at Weeks 3, 6, or 9 to the next highest dose level if blood pressure goal not achieved
  Interventions: Drug: losartan potassium
- Losartan potassium 0.7 to 1.4 mg/kg (Experimental): Open-label losartan at starting dose of 0.7 mg/kg/day with uptitration at Weeks 3, 6, or 9 to the next highest dose level if blood pressure goal not achieved
  Interventions: Drug: losartan potassium

INTERVENTIONS:
Drug: losartan potassium — losartan potassium, dry powder, to be suspended in liquid and given orally, once daily; doses will start at 0.1 mg/kg, 0.3 mg/kg, and 0.7 mg/kg, respectively, in the three study arms and can be escalated up to 1.4 mg/kg (maximum dose 100 mg) until target blood pressure is reached.
  Other Names: Cozaar

SUMMARY:
This study will explore the dose-response of losartan as well as the safety and tolerability in children from 6 months to 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participant is determined to be hypertensive

Exclusion Criteria:

* Participant has a history of severe or symptomatic hypertension
* Participant has history of heart failure, rhythm disturbance or cardiomyopathy, or obstructive valvular disease
* Participant has started taking hypertensive medications within the past 30 days
* Participant has a known sensitivity to losartan or history of angioneurotic edema

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2012-08-14 (Actual); Study Completion 2012-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Webb NJ, Wells TG, Shahinfar S, Massaad R, Dankner WM, Lam C, Santoro EP, McCrary Sisk C, Blaustein RO. A randomized, open-label, dose-response study of losartan in hypertensive children. Clin J Am Soc Nephrol. 2014 Aug 7;9(8):1441-8. doi: 10.2215/CJN.11111113. Epub 2014 May 29. PMID 24875194

RESULTS

PARTICIPANT FLOW:
Groups:
- Losartan Potassium 0.3 to 1.4 mg/kg: Open-label losartan at starting dose of 0.3 mg/kg/day with uptitration at Weeks 3, 6 or 9 to the next highest dose level if blood pressure goal not achieved
- Losartan Potassium 0.7 to 1.4 mg/kg: Open-label losartan at starting dose of 0.7 mg/kg/day with uptitration at Week 3, 6, or 9 to the next highest dose level if blood pressure goal not achieved
- Losartan Potassium-Extension: Participants who elected to enter extension; dose level of Losartan was that which was being administered at end of base study
Period: 12-week Base Study
Arm/Group | Losartan Potassium 0.1 to 1.4 mg/kg | Losartan Potassium 0.3 to 1.4 mg/kg | Losartan Potassium 0.7 to 1.4 mg/kg | Losartan Potassium-Extension
Started | 33 | 34 | 34 | 0
Completed | 31 | 34 | 32 | 0
Not Completed | 2 | 0 | 2 | 0
Not completed — Protocol-specific Criteria Met | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Period: Optional Extension
Arm/Group | Losartan Potassium 0.1 to 1.4 mg/kg | Losartan Potassium 0.3 to 1.4 mg/kg | Losartan Potassium 0.7 to 1.4 mg/kg | Losartan Potassium-Extension
Started | 0 | 0 | 0 | 90 (7 participants who completed base study opted not to enter extension)
Completed | 0 | 0 | 0 | 53
Not Completed | 0 | 0 | 0 | 37
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — End of Study | 0 | 0 | 0 | 11
Not completed — Protocol-specific criteria met | 0 | 0 | 0 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan Potassium 0.1 to 1.4 mg/kg | Losartan Potassium 0.3 to 1.4 mg/kg | Losartan Potassium 0.7 to 1.4 mg/kg | Total
Number analyzed (Participants) | 33 | 34 | 34 | 101
Age, Continuous [Mean (Standard Deviation); unit: Months] | 40.2 (24.4) | 45.0 (21.5) | 40.6 (21.2) | 42.0 (22.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 14 | 43
  Male | 20 | 18 | 20 | 58

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure
Description: Sitting blood pressure ([BP] or supine if child could not sit) was measured after the participant had been seated for 5 minutes with back supported, feet on the floor and right arm (or left arm if it was the customary side for BP measurement for the patient) supported at heart level. Systolic BP was determined by averaging 3 replicate measurements obtained at least 1 minute apart.
Time Frame: Baseline and Day 21
Population: Analysis performed using the Full Analysis Set defined as all randomized participants who had at least 1 dose of study drug, had baseline data, and had a post-treatment endpoint observation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan Potassium 0.1 to 1.4 mg/kg | Losartan Potassium 0.3 to 1.4 mg/kg | Losartan Potassium 0.7 to 1.4 mg/kg
Number analyzed (Participants) | 32 | 34 | 33
mmHg | -7.31 (12.53) | -7.65 (7.49) | -6.67 (7.86)
Statistical Analysis 1: Comparison: Losartan Potassium 0.1 to 1.4 mg/kg vs Losartan Potassium 0.3 to 1.4 mg/kg vs Losartan Potassium 0.7 to 1.4 mg/kg; Test type: Superiority or Other; p = 0.753, ANCOVA; Analysis of covariance (ANCOVA) model with terms for dose, weight (as a continuous covariate) and presence of co-morbidities/end organ damage; Slope = 1.22, 95% CI 2-sided [-6.45 to 8.90]

2. Secondary Outcome: Mean Change From Baseline in Diastolic Blood Pressure
Description: Sitting BP (or supine if child could not sit) was measured after the participant had been seated for 5 minutes with back supported, feet on the floor and right arm (or left arm if it was the customary side for BP measurement for the patient) supported at heart level. Diastolic BP was determined by averaging 3 replicate measurements obtained at least 1 minute apart.
Time Frame: Baseline and Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Losartan Potassium 0.1 to 1.4 mg/kg | Losartan Potassium 0.3 to 1.4 mg/kg | Losartan Potassium 0.7 to 1.4 mg/kg
Number analyzed (Participants) | 32 | 34 | 33
mmHg | -8.25 (11.76) | -5.15 (8.06) | -6.73 (8.59)
Statistical Analysis 1: Comparison: Losartan Potassium 0.1 to 1.4 mg/kg vs Losartan Potassium 0.3 to 1.4 mg/kg vs Losartan Potassium 0.7 to 1.4 mg/kg; Test type: Superiority or Other; p = 0.643, ANCOVA; [statistical method as in outcome 1, analysis 1]; Slope = 1.81, 95% CI 2-sided [-5.90 to 9.51]

3. Primary Outcome: Number of Participants Who Reported 1 or More Clinical and/or Laboratory Adverse Event(s)
Time Frame: up to 12 weeks (Base Study); up to 24 months (Extension)
Population: All Patients as Treated Population, which consisted of all randomized participants who received at least 1 dose of study drug. Adverse events for the base study were reported by the dose taken at the time of the event and not the study group to which they were randomly assigned. Adverse events for the study extension were reported as 1 arm.
Measure: Number; unit: Participants
Groups:
- Base Study-Losartan Potassium 0.1 mg/kg: Open-label Losartan 0.1 mg/kg/day
- Base Study-Losartan Potassium 0.3 mg/kg: Open-label Losartan 0.3 mg/kg/day
- Base Study-Losartan Potassium 0.7 mg/kg: Open-label Losartan 0.7 mg/kg/day
- Base Study-Losartan Potassium 1.4 mg/kg: Open-label losartan 1.4 mg/kg/day
- Extension-Losartan Potassium: Open-label losartan at dose of 0.1, .03, .07 or 1.4 mg/kg/day
Arm/Group | Base Study-Losartan Potassium 0.1 mg/kg | Base Study-Losartan Potassium 0.3 mg/kg | Base Study-Losartan Potassium 0.7 mg/kg | Base Study-Losartan Potassium 1.4 mg/kg | Extension-Losartan Potassium
Number analyzed (Participants) | 34 | 54 | 63 | 33 | 90
Participants
  Clinical Adverse Event | 21 | 30 | 36 | 22 | 75
  Laboratory Adverse Event | 1 | 1 | 0 | 0 | 5

4. Primary Outcome: Number of Participants Who Were Discontinued From Study Due to a Clinical and/or Laboratory Adverse Event
Time Frame: up to 12 weeks (Base Study); up to 24 months (Extension)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Base Study-Losartan Potassium 0.1 mg/kg | Base Study-Losartan Potassium 0.3 mg/kg | Base Study-Losartan Potassium 0.7 mg/kg | Base Study-Losartan Potassium 1.4 mg/kg | Extension-Losartan Potassium
Number analyzed (Participants) | 34 | 54 | 63 | 33 | 90
Participants
  Clinical Adverse Event | 0 | 0 | 0 | 0 | 1
  Laboratory Adverse Event | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 weeks (Base Study); up to 24 months (Extension)
Description: Serious and Non-serious adverse events are reported by the dose taken at the time of the event and not the study group to which they were randomly assigned. A participant may have reported a serious/adverse event when taking different dose levels and therefore may have been counted more than once.
Arm/Group | Base Study-Losartan Potassium 0.1 mg/kg/Day | Base Study-Losartan Potassium 0.3 mg/kg/Day | Base Study-Losartan Potassium 0.7 mg/kg/Day | Base Study-Losartan 1.4 mg/kg/Day | Extension-Losartan 0.1 mg/kg/Day | Extension-Losartan 0.3 mg/kg/Day | Extension-Losartan 0.7 mg/kg/Day | Extension-Losartan 1.4 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 3/34 | 2/54 | 2/63 | 0/33 | 3/15 | 5/28 | 2/31 | 5/42
Other Adverse Events (participants affected / at risk) | 15/34 | 22/54 | 23/63 | 17/33 | 12/15 | 20/28 | 20/31 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study-Losartan Potassium 0.1 mg/kg/Day (N=34) | Base Study-Losartan Potassium 0.3 mg/kg/Day (N=54) | Base Study-Losartan Potassium 0.7 mg/kg/Day (N=63) | Base Study-Losartan 1.4 mg/kg/Day (N=33) | Extension-Losartan 0.1 mg/kg/Day (N=15) | Extension-Losartan 0.3 mg/kg/Day (N=28) | Extension-Losartan 0.7 mg/kg/Day (N=31) | Extension-Losartan 1.4 mg/kg/Day (N=42)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study-Losartan Potassium 0.1 mg/kg/Day (N=34) | Base Study-Losartan Potassium 0.3 mg/kg/Day (N=54) | Base Study-Losartan Potassium 0.7 mg/kg/Day (N=63) | Base Study-Losartan 1.4 mg/kg/Day (N=33) | Extension-Losartan 0.1 mg/kg/Day (N=15) | Extension-Losartan 0.3 mg/kg/Day (N=28) | Extension-Losartan 0.7 mg/kg/Day (N=31) | Extension-Losartan 1.4 mg/kg/Day (N=42)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2) | 3 (4) | 3 (5) | 5 (5) | 6 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (7) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 3 (3) | 4 (6) | 3 (3) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 4 (10)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7) | 3 (3) | 2 (3) | 2 (3) | 4 (6) | 5 (6) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 5 (6) | 3 (3) | 2 (2) | 3 (3) | 3 (6) | 5 (13)
Rhinitis (Infections and infestations) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 5 (6)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (8) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (3) | 2 (2) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 3 (12) | 7 (13)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Lip and/or oral cavity cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 5 (9)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to the multicenter publication, or 24 months after completion of the study, whichever comes first, an investigator and/or his/her colleagues may publish the results for their study site independently. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.